CLINICAL TRIAL: NCT06377605
Title: The Efficacy of Thoracic Erector Spinae Plane Block For Perioperative Analgesia in Laparoscopic Bariatric Surgery for Super Obese Patients: Randomized Controlled Trial
Brief Title: The Efficacy of Thoracic Erector Spinae Plane Block For Perioperative Analgesia in Laparoscopic Bariatric Surgery for Super Obese Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amany Ahmed Eissa (Other)
Responsible Party: Sponsor-Investigator, Amany Ahmed Eissa, lecturer of anesthesia& ICU, Kasr El Aini Hospital
Organization: Kasr El Aini Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD-15-2024
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Erector Spinae Plane Block; Super Obese Patients; Bariatric Surgery
Keywords: super obese; ESPB; bariatric
MeSH Terms: interventions — Midazolam; Lidocaine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: randomized controlled trial- single blinded
Who Masked: Participant
Masking Description: Computer-generated sequence will be used for randomization and opaque envelopes will be used for concealment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector Spinae block . (Active Comparator): the block will be performed preoperatively with 1mg midazolam administration intravenous , and 5 cm lidocaine 1% infiltration at each side prior to the block .
  the patient will be placed in the lateral or sitting position . The block will be performed bilaterally by injecting 60 mL of 0.25% bupivacaine (30 mL into each side) [16] into the fascial plane between the deep surface of the Erector Spinae muscle and the transverse processes of the lumbar vertebrae laterally (at the most lateral part of the transverse process) and since it is a fascial plane block , the greater the volume of the local anaesthetic injected , the distribution will be better.
  Interventions: Procedure: ESPB; Drug: midazolam and lidocaine
- local anaesthetic infiltration (Active Comparator): : the participant will receive 5 ml bupivacaine infiltration to each trocar site (total of 25 ml 0.5 %) at the beginning of the operation.
  Interventions: Procedure: local anaesthetic infiltration; Drug: Bupivacain

INTERVENTIONS:
Procedure: ESPB — the target vertebral level ( T7 transverse process ) [8] in the lateral or sitting position and moved in approximately 3-cm lateral to the spinous process . The Erector Spinae muscle and transverse process will be then identified, and a blunted tip , 20-gauge, short bevel needle (Pajunk Sonoplex, Geisingen, Germany) will be advanced, using the in-plane approach, in cephalad-to-caudal direction, through the interfascial plane between the Erector Spinae and the underlying transverse process under strict aseptic precautions until the tip is deep to erector spinae muscle. The block will be performed bilaterally by injecting 60 mL of 0.25% bupivacaine (30 mL into each side) [16] into the fascial plane between the deep surface of the Erector Spinae muscle and the transverse processes of the lumbar vertebrae laterally (at the most lateral part of the transverse process) and since it is a fascial plane block , the greater the volume of the local anaesthetic injected ,
  Arms: Erector Spinae block .
Procedure: local anaesthetic infiltration — the participant will receive 5 ml bupivacaine infiltration to each trocar site (total of 25 ml 0.5 %) at the beginning of the operation.
  Arms: local anaesthetic infiltration
Drug: midazolam and lidocaine — midazolam administration intravenous , and 5 cm lidocaine 1% infiltration
  Arms: Erector Spinae block .
Drug: Bupivacain — bupivacaine infiltration
  Arms: local anaesthetic infiltration

SUMMARY:
The epidemic of overweight and obesity presents a major challenge to chronic disease prevention and health across the life course around the world. [1] Bariatric surgery has proved to be an efficient intervention in the management of obesity. As a result, the number of post-bariatric surgery patients in the population is growing [2].

Postoperative analgesia presents various challenges in vulnerable patient groups suffering from obesity. With the high potential risk of respiratory depression and postoperative pulmonary complications associated with opioid use, such as atelectasis and pneumonia, the availability of other pain management modalities is essential [14].

Ultrasound-guided erector spinae plane block (ESPB) is a regional anesthesia technique where local anesthetic agent is injected deep to the erector spinae muscle to fascial plane and allowed to diffuse caudally and cranially. It is supposed to provide both visceral and somatic abdominal analgesia [3].

ESPB is effective, easy to perform, and can be performed in a short time. [4] It has been shown efficacy in different conditions such as thoracic surgery, trauma, cardiac surgery, breast surgery, and abdominal surgery [5]. However, the main concern with the ESPB block is feasibility together with the potency of the block in challenging populations, such as patients suffering from obesity.

Peripheral nerve blocks in the obese may pose challenges, like difficulties in proper patient positioning and landmark identification. However, Ultrasound guidance may help overcome many difficulties in regional techniques. But as expected, targets are more deeply situated in obese patients and the ultrasound beams are attenuated as they travel a greater distance through tissue layers. Additionally, when crossing a tissue boundary, a portion is reflected back to the transducer creating artifacts like speckling and clutter which are particular problems in the obese patient. [15] Few studies examined the use of ESPB in bariatric surgery [3,6,7], all indicating potential benefits of the technique in terms of opioid sparing and pain control. To date, the efficacy of ESPB has not been examined in superobese patient.

So we aim to compare the perioperative analgesic effect of bilateral ultrasound-guided ESPB with controls, Local bupivacaine infiltration to the trocar sites, in super obese patients undergoing bariatric surgery We hypothesis that ESBP provides good applicable modality of perioperative analgesia for superobese patients undergoing bariatric surgeries.

DETAILED DESCRIPTION:
Following approval from Ethics and Research Committee of Anaesthesia Department, Faculty of Medicine, Cairo University; 60 patients fulfilling inclusion criteria will be included in this randomized prospective comparative trial.

A.preoperative:

History will be taken from all patients. Age and then American Society Anaesthesiologists' (ASA) score will be recorded.

Preoperatively patients' laboratory investigations as complete blood picture, coagulation profile, liver and renal functions will be recorded. General examination will be carried out with examination of the back to exclude infection at the injection site and anatomical deformities.

Baseline vital signs will be recorded including non-invasive measurement of systolic, mean, diastolic arterial pressures, and HR and oxygen saturation. After inserting an intravenous (IV) access, the patient will be pre-medicated with metoclopramide in a dose 0.1-0.2 mg/kg.

Patient will be randomly assigned into 1 of 2 groups according to the intervention used whether:

* Group A (30 patients): Erector Spinae block .
* Group B (30 patients): local anaesthetic infiltration. Upon arrival to O.R; perioperative monitoring including continuous Electro Cardio Gram (GE-Datex Ohmeda 5 leads ECG cable), pulse oximetry (GE- Datex Ohmeda finger SpO2 sensor), non-invasive arterial blood pressure (GE-Datex Ohmeda NIBP cuff) will be applied.

In group A, block will be performed by the primary investigator the the block will be performed preoperatively with 1mg midazolam administration intravenous , and 5 cm lidocaine 1% infiltration at each side prior to the block .

the patient will be placed in the lateral or sitting position . Then, the Erector Spinae block will be given by a high-frequency linear ultrasound transducer of Siemens acuson x300 3-5MHz ultrasound . It will be sagittally placed against the target vertebral level ( T7 transverse process ) [8] in the lateral or sitting position and moved in approximately 3-cm lateral to the spinous process . The Erector Spinae muscle and transverse process will be then identified, and a blunted tip , 20-gauge, short bevel needle (Pajunk Sonoplex, Geisingen, Germany) will be advanced, using the in-plane approach, in cephalad-to-caudal direction, through the interfascial plane between the Erector Spinae and the underlying transverse process under strict aseptic precautions until the tip is deep to erector spinae muscle, as evidenced by visible hydro-dissection below the muscle plane, and on injection of 5 ml normal saline to confirm the correct needle tip position. The block will be performed bilaterally by injecting 60 mL of 0.25% bupivacaine (30 mL into each side) [16] into the fascial plane between the deep surface of the Erector Spinae muscle and the transverse processes of the lumbar vertebrae laterally (at the most lateral part of the transverse process) and since it is a fascial plane block , the greater the volume of the local anaesthetic injected , the distribution will be better.

B.intraoperative:

Then, general anaesthesia will be induced in both groups . 1-2 μg/kg fentanyl based on lean body weight [3] with maximum dose of 200 μg and 2 mg/kg propofol will be given based on total body weight [3]. Tracheal intubation will be facilitated with 0.5 mg/kg atracurium based on ideal body weight [10].

In Group (B) Control group : the participant will receive 5 ml bupivacaine infiltration to each trocar site (total of 25 ml 0.5 %) at the beginning of the operation.

For both groups, Anaesthesia will be maintained using isoflurane in oxygen and air. Additional doses of 0.1 mg/kg atracurium will be administrated every 30 minutes. The surgical intervention will be then allowed 20 minutes after finishing the block procedure in group (A).

Pressure control volume guarantee ventilation will be adjusted to maintain normocapnia. Anesthesia will be maintained by using 1-1.5% isoflurane in a mixture of oxygen and air (50/50) and atracurium top ups at a dose of 0.1mg/kg every 30 minutes.

All participants will be given 1 gram of intravenous paracetamol with maximum dose of 4 gm every 24 hour Failed block ( increase in HR and mean arterial blood pressure (MABP)>20% from base line with skin incision) will be treated by 1ug /kg of fentanyl as top-up doses and increasing isoflurane concentration in case of inadequate response to fentanyl.

20 minute before the end of the surgery ketorolac 0.5mg/kg diluted in 100 ml of saline will be given intravenously After skin closure, inhalational anesthesia will be discontinued and reversal of muscle relaxation with atropine (0.02 mg/Kg) and neostigmine (0.05 mg/Kg) will be administered intravenous after return of patient's spontaneous breathing. Patients will then be transferred to post anesthesia care unit (PACU) for 60 min to complete recovery and monitoring.

At any time hypotension (defined as a decrease in mean arterial pressure (MAP) >20% from baseline value or systolic arterial pressure (SAP <100 mmHg) will be treated with 5 mg IV bolus ephedrine and repeated every 3 minutes until the hypotension resolved. Bradycardia (defined as a HR <40 beats per minute ) will be treated with atropine 0.5 mg IV.[11]

C.postoperative:

In the PACU; VAS will be assessed 15 min after extubation and when the score exceeds 3/10, rescue analgesia in the form of nalbuphine 0.1 mg/Kg with maximum dose of 30 mg every 24 hours will be given. Another dose of nalbuphine 0.1 mg/kg can be given in the PACU if the score still more than 3 after 30 min of the 1st dose.

After discharging from the PACU, the analgesic plan will be intravenous paracetamol one gram every 8 hours , ketorolac 0.5mg/kg/ 6 hours if VAS score > 3 and nalbuphine as second rescue analgesia 0.1 mg/kg /8 hours as long as the pain score is more than 3\10 ( reassessment to be done after 30 mins of administration of first rescue analgesia ) .

3. Measurement tools

* Patients characteristics including patient's age in years, weight in kilograms,BMI, gender, type of surgery.
* All hemodynamic parameters as blood pressure using non-invasive measurement, heart rate, oxygen saturation will be recorded at baseline , 5 mins after intubation ,every 10 min till the end of the surgery , immediately after extubation , 5 min after extubation , and every 10 mins in PACU for 30 min till the discharge of the patient .
* Failed blocks will be documented (patient requirement of consecutive rescue analgesia).
* the patients will be evaluated regarding the time to first demand to rescue analgesia postoperatively.

  * The pain will be assessed by the VAS score, It will be performed in the immediate post-operative period every 30 min for the first hour , 2 h, 4 h, 8h, 12h and 24 h. Breakthrough pain will be defined as VAS >3 at rest.
* Pain will be classified as mild (VAS 1-3), moderate (VAS 4-6), and severe (VAS 7-10) .
* Postoperative regular analgesia will be prescribed for all patients in the form of paracetamol every 8 hours. Rescue analgesia will be administered, if VAS is >3 at any time with IV ketorolac 0.5 mg/kg diluted in 100 ml normal saline and administered slowly every 6 hours .

Reassessment of VAS score will be done and if VAS is still > 3 the second rescue analgesic planned will be IV nalbuphine 0.1 mg/kg every 8 hours .

* The time interval between the first and the second rescue analgesia will be 30 minutes if VAS score remains persistently >3 .
* Time at which the patient start to ambulate in both groups will be recorded [12]
* PONV in first 24hr will be monitored and documented if occurred.

  * complications such as hematoma at the site of injection and local anesthetic toxicity will be documented .
  * Quality of recovery questionnaire.QoR15.

VI. Study outcomes

1. Primary outcome Total opioid consumption (morphine equivalent dose) in both groups in 24hr postoperative (including Intraoperative fentanyl , and postoperative nalluphine).
2. Secondary outcome(s)

   1. VAS score during first 24 hour postoperative
   2. Failure rate in performing the block
   3. Patient demographic data (age ,sex ,ASA classification ,BMI and type of surgery).
   4. Postoperative nausea and vomiting in first 24 hours.
   5. Time at which the patient start to ambulate in both groups
   6. Haemodynamic parameters (heartrate,Blood pressure) recorded intraoperative ,immediately postoperatively and in PAICU.
   7. Incidence of complications related to the block as infection or hematoma at the site of injection , local anaesthetic toxicity or pneumothorax .
   8. Time for first rescue analgesia in both groups.
   9. Quality of recovery questionnaire (QoR15) after 24hr from the end of the surgery

ELIGIBILITY:
Inclusion Criteria:

* Patient age >18 <60

  * Super Obese patients ; Body mass index(BMI) > 50 kg/m2
  * Both sexes
  * American Society of Anesthesiologists(ASA) physical status classes II and III
  * Patients scheduled for laparoscopic bariatric surgery i.e. sleeve gastrectomy and/or Roux-en-Y gastric bypass (RYGB)surgeries

Exclusion Criteria:

* • Refusal of regional block

  * Patients with neurological, psychological disorders or those lacking cooperation
  * Patients scheduled for concomitant laparoscopic cholecystectomy or paraumbilical hernia repair or those with history of previous bariatric surgery or obstructive sleep apnea
  * Patients with anatomic abnormalities at site of injection, skin lesions or wounds at site of proposed needle insertion.
  * Patients with bleeding disorders defined as (INR >1.4) and/ or (platelet count <100,000/µL)
  * Patients with hepatic disease e.g. liver cell failure or hepatic malignancy or hepatic enlargement.
  * Patients who are allergic to amide local anesthetics.
  * Cases converted to open surgery will also be excluded from the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption | 24 hours
  (morphine equivalent dose) in both groups in 24hr postoperative (including Intraoperative fentanyl , and postoperative nalluphine).

SECONDARY OUTCOMES:
VAS score during first 24 hour postoperative | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Ainy Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No